CLINICAL TRIAL: NCT01856439
Title: A Multicentre, Open-label Study to Determine the Long Term Safety, Tolerability and Efficacy of ProSavin in Patients With Bilateral, Idiopathic Parkinson's Disease.
Brief Title: Long Term Safety and Efficacy Study of ProSavin in Parkinson's Disease
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: As a result of termination of development of Prosavin, it is no longer possible for Sio to either commence or to continue any related clinical trials.
Sponsor: Axovant Sciences Ltd. (Industry)
Collaborators: Oxford BioMedica (Industry)
Responsible Party: Sponsor
Organization: Sio Gene Therapies (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PS1/001/09; 2009-017253-35 (EudraCT Number)
Record Dates: First submitted 2013-05-14; First posted 2013-05-17 (Estimated); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Parkinson's Disease
Keywords: ProSavin; Gene therapy
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Long term follow up (Other): Long term follow up of patient's who received ProSavin in previous study
  Interventions: Drug: ProSavin

INTERVENTIONS:
Drug: ProSavin — Long term follow up of patients who received ProSavin in a previous study

SUMMARY:
The study is designed to assess the long term tolerability of ProSavin and whether it is safe and efficacious in patients administered ProSavin from the PS1/001/07 study .

ELIGIBILITY:
Inclusion Criteria:

* must have met all inclusion criteria for study PS1/001/07
* willing to have L-DOPA dosage reduced/withdrawn at the discretion of the investigator at regular intervals to allow assessment of ProSavin in the absence of concomitant antiparkinsonian medication.
* affiliated with the French social security health care system (Patients enrolled in France only)
* signed and dated written informed consent obtained from the patient and/or the patient's legally acceptable representative, if applicable, in accordance with the local regulations
* must have been treated with ProSavin/Sham

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-05; Primary Completion 2021-11 (Actual); Study Completion 2022-04 (Actual)

PRIMARY OUTCOMES:
To assess the long term safety and tolerability of ProSavin | 10 years
  The number and severity of any adverse event

SECONDARY OUTCOMES:
Patients' responses to ProSavin administration | 10 years
  Assessed using Unified Parkinson's Disease Rating Score(UPDRS) Part III, evaluating percentage of time during waking day that patient is in the "off" state through patient diaries and activities of daily living using PDQ-39 at 36 months post administration.

CONTACTS AND LOCATIONS:
Overall Officials: Stephane Palfi, Professor, Principal Investigator — Henri Mondor University Hospital; Roger Barker, Dr, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (2):
- Henri Mondor Hospital, Paris, France
- Addenbrookes Hospital, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Palfi S, Gurruchaga JM, Ralph GS, Lepetit H, Lavisse S, Buttery PC, Watts C, Miskin J, Kelleher M, Deeley S, Iwamuro H, Lefaucheur JP, Thiriez C, Fenelon G, Lucas C, Brugieres P, Gabriel I, Abhay K, Drouot X, Tani N, Kas A, Ghaleh B, Le Corvoisier P, Dolphin P, Breen DP, Mason S, Guzman NV, Mazarakis ND, Radcliffe PA, Harrop R, Kingsman SM, Rascol O, Naylor S, Barker RA, Hantraye P, Remy P, Cesaro P, Mitrophanous KA. Long-term safety and tolerability of ProSavin, a lentiviral vector-based gene therapy for Parkinson's disease: a dose escalation, open-label, phase 1/2 trial. Lancet. 2014 Mar 29;383(9923):1138-46. doi: 10.1016/S0140-6736(13)61939-X. Epub 2014 Jan 10. PMID 24412048